CLINICAL TRIAL: NCT01022021
Title: Adequacy of Peripheral Blood Stem Cell Mobilization in Patients With Relapsed Lymphoma Treated With Bendamustine: A Pilot Project and a Proof of Concept Study
Brief Title: Peripheral Blood Stem Cell (PBSC) Mobilization in Patients With Relapsed Lymphoma Treated With Bendamustine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11908
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Lymphoma
Keywords: non-Hodgkin's lymphoma; autologous stem cell transplant
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rituximab (Active Comparator)
  Interventions: Drug: Rituximab
- bendamustine (Active Comparator): bendamustine, 90 mg/M2
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Rituximab — Day 1 - rituximab, 375 mg/M2 IV (drug dosage is based on body weight)
  Other Names: Rituxan
  Arms: rituximab
Drug: Bendamustine — Days 2 and 3 bendamustine, 90 mg/M2 IV over 30-60 minutes (drug dosage based on body weight)
  Other Names: Treanda
  Arms: bendamustine

SUMMARY:
Patients with certain types of cancer require treatment with very high doses of chemotherapy. A side effect of high chemotherapy doses is damage to the bone marrow where our blood and immune system cells are produced.

Stem cells (or progenitor cells) are the source of all blood cells. They are formed in the bone marrow (the spongy cavity in the center of large bones). The stem cells receive signals that direct them to become red cells, white cells or platelets. This happens before they are released into the blood stream. Stem cells circulating in the blood stream can be collected through a process called "apheresis" or "stem cell collection". The cells are then processed and frozen to preserve them. After chemotherapy has been given the stem cells are thawed and given back intravenously (IV: into the vein), like a blood transfusion. The stem cells in the collection will find their way back into the bone marrow space and, after a few days, will start to produce the blood and immune cells as they normally would. Having your own stem cells collected and returned to you later is called an "autologous transplant."

Non-Hodgkin's lymphoma is a disease in which malignant cancer cells form in the lymph system. Autologous stem cell transplantation is the standard of care for a chemo-sensitive relapse in patients with large cell lymphoma that has spread.

Bendamustine works by blocking the growth of cancer cells. It is used for the management of chronic lymphocytic leukemia and follicular lymphoma. Bendamustine in addition to rituximab (BR) is used in several trials in patients with lymphoma with encouraging results. Adequate peripheral blood stem cell (PBSC) collection is a pre-requisite for high dose therapy followed by cell transplantation in patients with relapsed lymphoma. Exposure to previous multiple chemotherapy and radiation treatment may lead to poor mobilization of PBSC. It is not known whether pre-treatment with bendamustine will adversely affect the process of PBSC mobilization and harvest. On the other hand, it is assumed that high dose alkylating agents like cyclophosphamide may actually help in breaking the bond between stem cells and the stromal cells in the marrow cavity and hence may lead to a better mobilization of PBSC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory C20+ non-Hodgkin's lymphoma (proven by biopsy, radiological findings or clinical exam) referred to BMT clinic of Kansas University Medical Center for consideration of autologous stem cell transplantation. No separate recruitment method or advertisement will be used to enroll patients.
* Age 18-70 years.

Exclusion Criteria:

* Pregnancy and nursing mother
* Karnofsky performance status less than 50%
* Life expectancy is severely limited by concomitant illness
* Uncontrolled arrhythmias or symptomatic cardiac disease precluding transplantation
* Symptomatic pulmonary disease precluding transplantation
* Serum creatinine greater than 1.8 mg/dL
* Serum bilirubin greater than 2 times upper limit of normal, SGPT greater than 3 times upper limit of normal
* Evidence of chronic active hepatitis or cirrhosis
* Unable to sign informed consent
* Allergy to Rituximab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of G-CSF induced PBSC mobilization after two cycles of rituximab and Bendamustine (BR) as salvage therapy in patients with relapsed non-Hodgkins lymphoma | Quarterly

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha Ganguly, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States